CLINICAL TRIAL: NCT00112398
Title: Randomised, Controlled Trial of Physician Prehospital Management of Severe Blunt Head Injury
Brief Title: Head Injury Retrieval Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment rate combined with a high rate of patients dropping in to the treatment group from standard care
Sponsor: CareFlight (Other)
Collaborators: NSW Motor Accident Authority (Unknown)
Responsible Party: Principal Investigator, Alan Garner, Medical Director, CareFlight
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIRT1
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Head Injuries, Closed
Keywords: Head injuries; Prehospital; Advanced Interventions
MeSH Terms: conditions — Head Injuries, Closed; Craniocerebral Trauma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard (paramedic) prehospital care (Active Comparator)
  Interventions: Procedure: Extended interventions by advanced level prehospital providers
- Physician prehospital care (Experimental)
  Interventions: Procedure: Extended interventions by advanced level prehospital providers

INTERVENTIONS:
Procedure: Extended interventions by advanced level prehospital providers — may include rapid sequence intubation (RSI) airway management, blood transfusions, surgical procedures, etc.

SUMMARY:
The study hypothesis is that advanced interventions as provided by a physician at an accident scene will decrease the death rate and the rate of severe disability in survivors of severe head injury. Extended interventions by advanced level prehospital providers may include rapid sequence intubation (RSI) airway management, blood transfusions, surgical procedures, etc.

DETAILED DESCRIPTION:
A randomised, controlled trial examining prehospital management of persons with severe blunt head injury, in the Sydney region. Treatments examined will be the current system consisting principally of paramedic management (standard care) compared with management by a retrieval team lead by a consultant anaesthetist, emergency physician or intensive care specialist. Patients for inclusion in the study will be identified by a paramedic screening all "000" calls to the ambulance service and identifying persons likely to have severe head injury. The principal outcome measure will be their degree of disability measured at 6 months post injury.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma Scale score of 3 to 8 due to blunt trauma as measured at the accident scene by the first prehospital team to arrive at the site.

Exclusion Criteria:

* Penetrating trauma
* Age less than 16 years
* No more than 5 casualties at the scene

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2005-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale Score | Six months post injury

SECONDARY OUTCOMES:
Length of hospital and intensive care unit stays | At hospital discharge
30 day survival and survival to discharge from the acute care hospital | At hospital discharge and 30 days
Extended Glasgow Outcome Scale Score | Six months post injury
Disability Rating scale | Six months post injury

CONTACTS AND LOCATIONS:
Overall Officials: Alan A Garner, FACEM, Principal Investigator — CareFlight
Locations (1):
- CareFlight, PO Box 159, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Garner AA, Mann KP, Fearnside M, Poynter E, Gebski V. The Head Injury Retrieval Trial (HIRT): a single-centre randomised controlled trial of physician prehospital management of severe blunt head injury compared with management by paramedics only. Emerg Med J. 2015 Nov;32(11):869-75. doi: 10.1136/emermed-2014-204390. Epub 2015 Mar 20. PMID 25795741
- [Derived] Garner AA, Fearnside M, Gebski V. The study protocol for the Head Injury Retrieval Trial (HIRT): a single centre randomised controlled trial of physician prehospital management of severe blunt head injury compared with management by paramedics. Scand J Trauma Resusc Emerg Med. 2013 Sep 14;21:69. doi: 10.1186/1757-7241-21-69. PMID 24034628